CLINICAL TRIAL: NCT05375916
Title: Comparison of Short-term Sustained-release Opioid With Immediate-release Opioid for Acute Pain Management Following Open Abdominal Urologic Surgeries
Brief Title: Comparison of Short-term Sustained-release Opioid in Open Abdominal Urologic Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00118895
Record Dates: First submitted 2022-04-27; First posted 2022-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Pain, Acute; Opioid Use
Keywords: Postoperative pain; Opioid; Sustained-release opioid
MeSH Terms: conditions — Acute Pain; Pain, Postoperative | interventions — Hydromorphone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sustained-release opioid (Experimental): 3mg of sustained-release hydromorphone three times a day
  Interventions: Drug: Hydromorphone
- Short-acting opioid (Active Comparator): 1-4 mg of short-acting hydromorphone 2-4 times a day as needed
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Hydromorphone — Sustained-release hydromorphone is a long-acting preparation opioid

SUMMARY:
The advantage of slow-release opioid allows for less fluctuation in drug (pain killer) levels in the blood and an extended period within the effective range for pain relief. The slow-release opioids have been preferred over the short-acting opioids because of the longer duration of action, which lessens the frequency and severity of end-of-dose pain.

Herein, the investigators propose the use of low dose slow-release opioid formulation offers better pain control in the first 48 hours post-operatively in open abdominal urologic surgeries.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, controlled trial looking at all adult patients undergoing open abdominal urologic surgeries. After assessing the inclusion/exclusion criteria, the patients will be randomized into one of two groups:

Group 1: Sustained-release (long-acting) opioid on a regular basis for 2 days with immediate-release (short-acting) opioid available on an 'as required' basis

Group 2: Immediate-release (short-acting) opioid on an 'as required' basis only.

All patients will have a general anesthetic at the discretion of the anesthesiologist in the operating room and intravenous opioid will be administered in accordance with the anesthesiologists' discretion.

Pain score and analgesic consumption are the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing open abdominal urologic surgeries
* ASA 1-3

Exclusion Criteria:

* Patient refusal
* history of chronic pain
* allergy to hydromorphone
* cannot swallow tablets

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Time to Mobilization | Time to mobilize postoperatively up to 5 days
  Ability to walk from bed to chair

SECONDARY OUTCOMES:
Opioid consumption of hydromorphone | Postoperatively in recovery, 24 hours, 48 hours and 72 hours postoperatively
  Consumption of hydromorphone
Pain score | postoperatively day 1, 2, 3
  Pain score using visual analogue scale 0-100

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada